CLINICAL TRIAL: NCT06772129
Title: The Effect of Aromatherapy on Delirium in Critically Elderly Patients Undergoing Fracture Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Senay Gokdemir (Other)
Responsible Party: Sponsor-Investigator, Senay Gokdemir, specialist nurse, Necmettin Erbakan University
Organization: Necmettin Erbakan University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SGokdemir
Record Dates: First submitted 2025-01-04; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Delirium - Postoperative
MeSH Terms: conditions — Emergence Delirium | interventions — Aromatherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aromatherapy group (Active Comparator): The intervention to be performed in addition to routine care is to apply 0.3ml lavender oil to the aromatherapy necklace and leave it in an area 30 cm away from the patient's bed.
  Interventions: Other: Aromatherapy
- control group (No Intervention): While normal care and treatment in intensive care will continue to be applied to this group, necessary measurements will be taken and recorded.

INTERVENTIONS:
Other: Aromatherapy — Studies have been reviewed and no lavender aromatherapy has been found to be used for delirium.
  Arms: aromatherapy group

SUMMARY:
The aim of this quasi-experimental study was to examine the effect of lavender aromatherapy on delirium in patients who underwent fracture surgery, were in intensive care, and were over 60 years old.

The main question of the study was, does lavender aromatherapy affect delirium scale scores? In order to examine the effect of lavender oil on delirium, the researcher will provide routine care to one group and apply aromatherapy to the other group.

Both groups will be evaluated by the researcher at eight-hour intervals with the Nu-DESC delirium screening scale and the results will be compared.

DETAILED DESCRIPTION:
The American Nurses Association has defined delirium as "acute, serious, and often preventable conditions that are usually accompanied by confusion, dehydration, or attacks on some system followed by confusion and a distressing course of life". The incidence of delirium in the postoperative period is quite high and delirium has been associated with longer intensive care unit or hospital stays, higher hospital costs, and increased mortality. Delirium is especially risky in elderly and critically ill patients. Although postoperative delirium is tried to be treated using medication, nonpharmacological prevention methods are considered the most important part of the treatment. One of these methods is aromatherapy and has recently been widely used in nursing research. The smell of waste caused by patients' sweating, urinary and fecal incontinence, bleeding, and antiseptics such as povidone iodide, chlorhexidine, alcohol, and other drugs used during the treatment process creates a hospital-specific odor. Hospital odor is also associated with poor perception of treatment and care. It is thought that it would be beneficial to put an aromatic essential oil such as lavender oil in the environment. The positive effects of aromatherapy with lavender oil on anxiety, stress, pain, sleep quality, nausea and vomiting, as well as its sedative, emotionally calming, antiseptic, analgesic and antispasmodic properties have been demonstrated by studies. Essential oils are considered safe to use because they have minimal side effects. Postoperative delirium is a common complication following hip fracture surgery in the elderly. It has been observed that studies on the development of delirium in the intensive care unit were mostly conducted with patients who underwent cardiovascular surgery. This study will be carried out to determine how lavender oil aromatherapy left in the environment to prevent delirium, which can have serious consequences in the elderly with postoperative fractures, affects delirium scores.

ELIGIBILITY:
Inclusion Criteria:

* Having had surgery for a fracture and being treated in the ICU
* Being 60 years of age or older
* Having a first measured Nu-Desc score of less than 2
* Having a Glasgow coma scale score of >13
* Being able to speak and understand Turkish

Exclusion Criteria:

* Having trouble smelling
* Being intubated
* Having asthma, COPD or any respiratory disorder
* Having been previously diagnosed with delirium
* Having other cognitive disorders such as Alzheimer's or dementia
* The patient needs to be physically restrained.
* Having multiple fractures.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
There is a difference between the delirium scores of aromatherapy and control elderly intensive care patients who have undergone fracture surgery. | The Nu-DESC score will be measured and recorded at 8-hour intervals for 24 hours after surgery.
  The Nu-DESC scale will be used to diagnose delirium. The Nu-DESC is an observational five-item scale that can be completed quickly. Symptoms are graded from 0 to 2 based on the presence and intensity of each symptom. Delirium may be considered if the patient's total score is 2 or higher.

CONTACTS AND LOCATIONS:
Overall Officials: Saide Faydalı, Associate Professor, Study Director — Necmettin Erbakan University, Faculty of Nursing

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Mosk CA, Mus M, Vroemen JP, van der Ploeg T, Vos DI, Elmans LH, van der Laan L. Dementia and delirium, the outcomes in elderly hip fracture patients. Clin Interv Aging. 2017 Mar 10;12:421-430. doi: 10.2147/CIA.S115945. eCollection 2017. PMID 28331300
- [Result] French J, Weber T, Ge B, Litofsky NS. Postoperative Delirium in Patients After Brain Tumor Surgery. World Neurosurg. 2021 Nov;155:e472-e479. doi: 10.1016/j.wneu.2021.08.089. Epub 2021 Aug 26. PMID 34455093
- [Result] Askarkafi F, Rayyani M, Dehghan M. The Effect of Massage With and Without Aromatic Oil on Delirium After Open-Heart Surgery: A Randomized Controlled Trial. J Chiropr Med. 2020 Mar;19(1):49-57. doi: 10.1016/j.jcm.2019.08.001. Epub 2020 Sep 3. PMID 33192191
- See also: American Delirium Society — https://americandeliriumsociety.org/
- See also: American Nursing Association — https://www.nursingworld.org/practice-policy/work-environment/health-safety/delirium/